CLINICAL TRIAL: NCT02552719
Title: Validation of the German Version of the Injustice Experience Questionnaire (IEQ) in 6 Pain Centers
Brief Title: Validation of the German Version of the Injustice Experience Questionnaire
Acronym: GIEVA
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Kantonsspital Baden (Other); Deutsches Rotes Kreuz DRK-Blutspendedienst Baden-Wurttemberg-Hessen (Other); Cantonal Hospital of St. Gallen (Other); University Hospital, Saarland (Other); Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: IEQ2015; SNCTP000000442 (Registry Identifier: kofam)
Record Dates: First submitted 2015-08-28; First posted 2015-09-17 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Validation Studies
Keywords: Injustice Experience; Questionnaire; Validation; German translation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Purpose of the study is the validation of the German version of the Injustice Experience Questionnaire.

Pretest: Participants were informed about the aims of the study and fill in a consent form. They filled in a paper version of the German translation of the Injustice Experience Questionnaire. In a structured interview patients were asked if there were any items difficult to understand, unacceptable or offending them. Subsequently they had to answer questions about the content and meaning of the IEQ-items.

Validation Study: Participants were informed about the aims of the study and filled in a consent form. By e-mail they received an access link to the online survey. The questionnaires of the survey could be filled in at home. The survey could be interrupted and terminated later. About 20 minutes were needed to answer the 80 questions of the survey. All data was saved anonymously during the survey.

DETAILED DESCRIPTION:
Pretest: Participants were informed about the aims of the study and filled in a consent form. A paper version of the German translation of the Injustice Experience Questionnaire was completed in presence of the interviewer. The structure of the standardized interview followed the recommendations for pretesting transcultural translations of questionnaires. Patients were asked if there were any items difficult to understand, unacceptable or offending them. Subsequently they had to answer questions about the content and meaning of the IEQ-items. The interviewer asked all questions and entered the responses. All data were directly stored in a MySQL database at a Swiss commercial web-server (www.scientific-affairs.ch).

Validation Study: Participants are informed about the aims of the study and fill in a consent sheet. By e-mail they receive an access link to the online survey which can be completed at home. The survey includes the following questionnaires: Injustice Experience Questionnaire (IEQ), Depression subscale of the Depression, Anxiety and Stress Scale (DASS), Tampa Scale for Kinesiophobia (TSK), McGill Pain Questionnaire (MPQ), Pain Catastrophizing Scale (PCS), Pain Disability Index (PDI) and part concerning causes of pain of the German Pain Questionnaire (DSF). About 20 minutes is needed to answer the 80 questions of the survey. After completing the survey participant can choose if they would like to be informed about the results of the filled in questionnaires. All data is saved anonymously during the survey and stored in a MySQL database at a Swiss commercial web-server (www.scientific-affairs.ch).

ELIGIBILITY:
Inclusion Criteria:

* pain (face, head or rest of the body)
* good competence of German language
* internet access
* being able to fill in a web-based survey
* adults

Exclusion Criteria:

* disuse / dependency on medication / drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pain patients
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of patients' confirmative responses related to the 12 IEQ-items in a questionnaire concerning 1) comprehensiveness, 2) acceptance, 3) offensiveness | 10 months
  patients answered if the IEQ-items were
  1. difficult to understand (yes/no)
  2. unacceptable (yes/no)
  3. offensive (yes/no)
Percentage of non-confirmative responses of two raters about the patients' considerations about 1) the meaning of IEQ-items, 2) the chosen response option | 10 months
  two raters judged if the patients' considerations about
  1. the meaning of the IEQ-items was understood (yes/no)
  2. the chosen response option was plausible (yes/no)
Correlations between the IEQ score and the scores of the MPQ, DASS_D, TSK, PCS, PDI | 7 months
  Correlations between the IEQ score and the scores of the MPQ, DASS_D, TSK, PCS, PDI are calculated and compared with the corresponding values English validation study.
Number of factors as the result of a factor analysis of the IEQ-items | 7 months
  Correspondence of the number of factors and the assigned items (as the result of a factor analysis) between the English and the German validation study

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Ettlin, MD, DMD, Principal Investigator — University of Zurich
Locations (6):
- Germany (2):
  - DRK Schmerz-Zentrum Mainz, Mainz, Rhineland-Palatinate
  - Schmerzambulanz der Klinik für Anästhesiologie, Intensivmedizin und Schmerztherapie, Universitätsklinikum des Saarlandes, Homburg, Saarland
- Switzerland (4):
  - ANNR Rehaclinic, Baden, Canton of Aargau
  - Zentrum für Schmerzmedizin, Schweizer Paraplegiker-Zentrum Nottwil, Nottwil, Canton of Lucerne
  - Kantonsspital St. Gallen, Schmerzzentrum, Sankt Gallen, Canton of St. Gallen
  - University of Zurich, Center of Dental Medicine, Zurich

REFERENCES:
- [Background] Sullivan MJ, Adams H, Horan S, Maher D, Boland D, Gross R. The role of perceived injustice in the experience of chronic pain and disability: scale development and validation. J Occup Rehabil. 2008 Sep;18(3):249-61. doi: 10.1007/s10926-008-9140-5. Epub 2008 Jun 7. PMID 18536983
- [Background] Stein C, Mendl G. The German counterpart to McGill Pain Questionnaire. Pain. 1988 Feb;32(2):251-255. doi: 10.1016/0304-3959(88)90074-7. PMID 3362561
- [Background] Sullivan, Michael J. L., Bishop SR, Pivik J. The Pain Catastrophizing Scale: Development and validation. Psychological Assessment 1995;7(4):524-532
- [Background] Meyer K, Sprott H, Mannion AF. Cross-cultural adaptation, reliability, and validity of the German version of the Pain Catastrophizing Scale. J Psychosom Res. 2008 May;64(5):469-78. doi: 10.1016/j.jpsychores.2007.12.004. PMID 18440399
- [Background] Kori S, Miller R, Todd D. Kinesiophobia: a new view of chronic pain behavior. Pain Management 1990:35-43
- [Background] Nigpur K, Russu AC. Fear of movement/(re)injury in chronic pain: Preliminary validation of a German version of the Tampa Scale for Kinesiophobia. European Journal of Pain 2009(13 (Supplement 1)):S239.
- [Background] Pollard CA. Preliminary validity study of the pain disability index. Percept Mot Skills. 1984 Dec;59(3):974. doi: 10.2466/pms.1984.59.3.974. No abstract available. PMID 6240632
- [Background] Dillmann U, Nilges P, Saile H, Gerbershagen HU. [Assessing disability in chronic pain patients.]. Schmerz. 1994 Jun;8(2):100-10. doi: 10.1007/BF02530415. German. PMID 18415443
- [Background] Melzack R. The McGill Pain Questionnaire: major properties and scoring methods. Pain. 1975 Sep;1(3):277-299. doi: 10.1016/0304-3959(75)90044-5. PMID 1235985